CLINICAL TRIAL: NCT01754974
Title: A Double-Blinded, Randomized Control Study Evaluating the Efficacy and Safety of Peginterferon Lambda-1a Compared to Peginterferon Alfa-2a, Each in Combination With Ribavirin, in the Treatment of Naive Genotype 1 Chronic Hepatitis C Subjects
Brief Title: Safety and Efficacy Study of Peginterferon Lambda-1a vs. Peginterferon Alfa-2a, Plus Ribavirin in Subjects With Genotype 1 Hepatitis C
Acronym: BASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI452-033; 2012-003508-11 (EudraCT Number)
Record Dates: First submitted 2012-12-19; First posted 2012-12-21 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2013-12

CONDITIONS: Hepatitis C Virus (HCV)
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon Lambda-1a + Ribavirin (Experimental): Peginterferon Lambda-1a 180 μg solution for subcutaneous (sc) injection once weekly and Ribavirin 1000 or 1200 mg based on weight tablet by mouth twice daily for 48 weeks
  Interventions: Biological: Peginterferon Lambda-1a; Drug: Ribavirin
- Peginterferon alfa-2a + Ribavirin (Active Comparator): Peginterferon alfa-2a 180 μg solution for subcutaneous (sc) injection once weekly and Ribavirin 1000 or 1200 mg based on weight tablet by mouth twice daily for 48 weeks
  Interventions: Drug: Ribavirin; Biological: Peginterferon alfa-2a

INTERVENTIONS:
Biological: Peginterferon Lambda-1a
  Other Names: BMS-914143
  Arms: Peginterferon Lambda-1a + Ribavirin
Drug: Ribavirin
  Other Names: Ribasphere
Biological: Peginterferon alfa-2a
  Other Names: Pegasys
  Arms: Peginterferon alfa-2a + Ribavirin

SUMMARY:
The purpose of this study is to determine if 48 weeks of therapy with Peginterferon Lambda plus Ribavirin is effective and safe for a treatment of chronic hepatitis C (CHC) compared to therapy with Peginterferon alfa-2a plus Ribavirin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hepatitis C, Genotype 1
* HCV RNA ≥100,000 IU/mL at screening
* Liver biopsy documenting no cirrhosis (within prior 3 years). Where approved for staging of liver disease, non-invasive imaging may be used to assess the extent of liver disease
* Naïve to prior anti-HCV therapy

Exclusion Criteria:

* Infected with HCV other than Genotype 1
* Positive Hepatitis B Surface Antigen (HBsAg), or Human Immunodeficiency Virus (HIV)-1/HIV-2 antibody at screening
* Evidence of liver disease other than HCV
* Active substance abuse
* Use of hematologic growth factors within 90 days prior to study randomization
* Evidence of history of cirrhosis based on radiologic criteria or biopsy results and clinical criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who develop treatment emergent cytopenic abnormalities (anemia as defined by Hb < 10 g/dL, and/or neutropenia as defined by ANC < 750 mm3 and/or thrombocytopenia as defined by platelets < 50,000 mm3) in treatment-naive subjects | Up to 48 weeks of treatment
  * ANC = Absolute Neutrophil Count
  * Hb = Hemoglobin

SECONDARY OUTCOMES:
Proportion of subjects with Sustained Virologic Response at Post-Treatment Follow-up Week 24 (SVR24), defined as Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) < Lower Limit of Quantitation of Assay (LLOQ) | At Post-Treatment Follow-up Week 24
Proportion of subjects with Rapid Virologic Response (RVR) (HCV RNA not detected) | On treatment Week 4 (of an up to 48-week treatment period)
Proportion of subjects with on-treatment Serious Adverse Events (SAEs) through end of treatment | Up to 48 weeks of treatment
Proportion of subjects with dose reductions through end of treatment | Up to 48 weeks of treatment
Proportion of subjects who discontinue due to Adverse Events (AEs) through end of treatment | Up to 48 weeks of treatment
Proportion of subjects with on-treatment Interferon (IFN)-associated symptoms as determined by adverse event reporting | Up to 48 weeks of treatment
  On-treatment IFN-associated symptoms are:
  * Flu-like symptoms (as defined by pyrexia or chills or pain)
  * Musculoskeletal symptoms (as defined by arthralgia or myalgia or back pain)
  * Neurological symptoms (headache or dizziness)
  * Constitutional symptoms (fatigue or asthenia)
  * Psychiatric symptoms (depression or irritability or insomnia)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (14):
- Czechia (3):
  - Local Institution, Hradec Králové
  - Local Institution, Prague
  - Local Institution, Ústí nad Labem
- Mexico (4):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Distrito Federal, Mexico City
  - Local Institution, Mexico City, Mexico City
  - Local Institution, México, State of Mexico
- South Korea (7):
  - Local Institution, Chungcheongnam-do
  - Local Institution, Daegu
  - Local Institution, Gangwon-do
  - Local Institution, Gyeonggi-do
  - Local Institution, Gyeongsangnam-do
  - Local Institution, Incheon
  - Local Institution, Seoul

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx